CLINICAL TRIAL: NCT06570577
Title: The Opioid Sparing Effect of an Inter-semispinalis Plane Block on Postoperative Pain Control in Posterior Cervical Spine Surgery
Brief Title: Opioid Sparing Effect of an ISP Nerve Block on Post-Op Pain Control in Posterior Cervical Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Eman Nada, Chief of Regional Anesthesia, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2024-00227
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative
Keywords: cervical fusion; opioids
MeSH Terms: conditions — Pain, Postoperative; Klippel-Feil Syndrome | interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: This is a randomized, blinded, 2-arm study of 60 participants. Two groups of 30 patients will be randomized to either 1) Routine pain management or 2) Inter-semispinalis Plane (ISP) Block plus Routine Pain Management.
Who Masked: Participant
Masking Description: Participants will be randomized using REDCap software. If the participant is randomized to the ISP Block group, it will be completed after the participant has been administered General Anesthesia and prior to surgery start.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Pain Management (Active Comparator): Routine Pain Management will include standard of care pharmacological management, by using patient-controlled opioid analgesia, oral acetaminophen, intravenous Ketorolac (Toradol), and Gabapentin. As needed (PRN), Intravenous hydromorphone will be given for breakthrough pain.
  Interventions: Drug: Opioids
- Routine Pain Management plus an Inter-semispinalis Plane Block (Experimental): Routine Pain Management, as described above, plus and ISP Block. After general anesthesia has begun, in the operating room, and the patient is moved to the prone position, before surgery start, those patients who are randomized to the block group, will receive a bilateral ISP nerve block in the back of the neck under ultrasound guidance, by a qualified, experienced Anesthesiologist.
  Under complete aseptic technique using an ultrasound guidance, 20 ml of Bupivacaine 0.25 % with 2 mg of Dexamethasone will be injected between two muscles in the back of the neck, bilaterally, to block the nerves that run in this plane.
  Once the block is completed, the surgical procedure will proceed as usual.
  Interventions: Procedure: Inter-semispinalis Plane Block

INTERVENTIONS:
Procedure: Inter-semispinalis Plane Block — A nerve block targeting the dorsal rami of the cervical spinal nerves can help alleviate postoperative incisional pain.
  Other Names: ISP nerve block
  Arms: Routine Pain Management plus an Inter-semispinalis Plane Block
Drug: Opioids — Routine Pain Management
  Other Names: Pharmacologic pain management
  Arms: Routine Pain Management

SUMMARY:
Participants who have a surgical procedure called Posterior Cervical (neck) Spine Surgery will normally need pain medication to relieve post operative pain. This usually includes opioid medications. In this study, the consented participant may receive a nerve block procedure, in addition to the pain relieving medication. There is a fifty-fifty chance to receive the nerve block. The goal is to see if the nerve block group needs less opioid medication, has lower pain scores and is discharged from the hospital sooner.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the opioid-sparing effect of the use of an Inter-semispinalis plane (ISP) block after posterior cervical spine surgery.

Posterior cervical fusion (PCF) is a painful procedure that often requires the use of high doses of opioids to minimize postoperative pain. Uncontrolled pain can result in a delay in recovery and discharge. Additionally, high doses of opioids carry the risk of opioid dependence, and other side effects, include nausea, vomiting, sedation, and, in rare cases, respiratory depression. For all of the above reasons, reducing the use of opioids is of utmost importance.

Nerve blocks are one alternative to opioid use. The ISP block is a procedure described in 2017; it is a relatively simple procedure that entails injecting local anesthetic between two muscles in the back of the neck, bilaterally, to block the nerves that run in this plane. It is done under ultrasound guidance and, although a limited number of studies have shown promise, more data on its safety and efficacy are needed. The addition of Dexamethasone to local anesthetics, in nerve blocks, resulted in significant prolongation of the analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Having Posterior Cervical Spine Surgery from C2 - C7, which may extend to the upper thoracic vertebrae, inclusive to T3.
* Capacity to provide informed consent

Exclusion Criteria:

* Fusion and decompression due to trauma
* Emergent procedures
* Patient is on a medication-assisted treatment, e.g., buprenorphine, naltrexone or methadone.
* There is an infection near or in the area of neck where the block will be placed.
* The patient is having a complicated surgery or a revision surgery
* Female patient with a positive pregnancy test on the day of surgery (hospital standard-of-care).
* Patient has Diabetes
* Patients who have had a prior adverse reaction to bupivacaine or dexamethasone
* Patients with Glucose-6-phosphate dehydrogenase deficiency or congenital or idiopathic methemoglobinemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Lower opioid use | 48 hours post Post-Anaesthesia Care Unit (PACU) arrival time
  Comparison of the reduction in Morphine Milligram Equivalent (MME) dose of opioids consumed between the control group versus the nerve block group.

SECONDARY OUTCOMES:
Lower opioid use. | MME use will be recorded from the patient's Anesthesia induction time until the patient's PACU arrival time. This will be the intra-operative period, which may last several hours, but not expected to exceed eight hours.
  MME from anesthesia induction time until PACU arrival time.
Lower opioid use | 24 hours after PACU arrival time
  MME for the 24 hours after PACU arrival time
Pain Scores | 48 hours after PACU arrival time
  Using a Numeric Rating Scale (NRS), pain scores will be obtained at specified times and then compared between the two groups. Participants will be asked to rate their pain on a scale from 0 - 10, where zero represents 'no pain at all' and 10 represents 'the worst pain ever possible'.
Length of hospital stay | The patient's EMR will record the date and time of admission, as well as, the date and time of discharge. This will be quantified by the REDCap software being used for this study, and is not expected to exceed four days.
  The length of hospital stay will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Nada, MBBCH, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No